CLINICAL TRIAL: NCT06598813
Title: Pediatric Headche Assessment Comparing PedMidas and HIT 6 Questionnaires
Brief Title: Pediatric Headche Assessment Using HIT 6
Status: Completed | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Jacob.genizi, Pediatric Neurologist, Bnai Zion Medical Center
Other Study IDs: BNZ187-22
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Headache Disorders, Primary
Keywords: HEADACHE; MIGRAINE; assessment; PEDMIDAS; HIT 6
MeSH Terms: conditions — Headache Disorders, Primary; Headache; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with haeadche: Children reporting headache for at least 3 month

SUMMARY:
The study is a prospective cohort study. The study population will include 100 children aged 6-18 years suffering from headaches who visited the Pediatric Neurology Clinic at Bnai Zion Medical Center and completed both the PED-MIDAS and HIT-6 questionnaires, starting from November 2022 until the end of the study period. Data will be collected from medical records and from the two questionnaires completed by the children during their clinic visit.

DETAILED DESCRIPTION:
Abstarct Background: Headache is one of the most common complaints in children and adolescents and is a leading cause of functional impairment in teenagers and young adults. The most common primary headaches being migraine and tension-type headache. Headaches negatively impact children's lives in various ways, with the effect varying according to the severity of the pain, the duration of the attack, and the response to treatment. To assess the degree of impact of headaches on daily functioning, the PED-MIDAS questionnaire was developed, tested, and validated in children aged 4-18 years, however, children often face difficulties in completing the questionnaire. The HIT-6 questionnaire, on the other hand, is user friendly however is validated only for adults.

Research Objectives: To compare the PED-MIDAS and HIT-6 questionnaires in their ability to assess the degree of impact of headaches on daily functioning.

Research Methods: The study is a prospective cohort study. The study population will include 100 children aged 6-18 years suffering from headaches who visited the Pediatric Neurology Clinic at Bnai Zion Medical Center and completed both the PED-MIDAS and HIT-6 questionnaires, starting from November 2022 until the end of the study period. Data will be collected from medical records and from the two questionnaires completed by the children during their clinic visit.

Research Importance: Children often struggle with completing the PED-MIDAS questionnaire because it requires them to recall the number of days their functioning was impaired over the three months prior to completing the questionnaire. This may lead to inaccurate completion and, consequently, an assessment that does not reflect the true impact. This created the need to compare the PED-MIDAS with the HIT-6 and examine whether it can serve as a better alternative.

ELIGIBILITY:
Inclusion Criteria:

* Chldern age 6-18 years with headache for at least 3 months.
* Children able to fill the questionnaire

Exclusion Criteria:

* Children with shoreter headaches.
* Children who are not able to fill the questionnaire

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with headache
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Hit 6 questionnaire | Once
  The hit 6 headache levels compered to the Pedmidas levels

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Cemter, Haif, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stewart WF, Lipton RB, Kolodner KB, Sawyer J, Lee C, Liberman JN. Validity of the Migraine Disability Assessment (MIDAS) score in comparison to a diary-based measure in a population sample of migraine sufferers. Pain. 2000 Oct;88(1):41-52. doi: 10.1016/S0304-3959(00)00305-5. PMID 11098098
- [Background] Stewart WF, Lipton RB, Dowson AJ, Sawyer J. Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability. Neurology. 2001;56(6 Suppl 1):S20-8. doi: 10.1212/wnl.56.suppl_1.s20. PMID 11294956
- [Background] Heyer GL, Perkins SQ, Rose SC, Aylward SC, Lee JM. Comparing patient and parent recall of 90-day and 30-day migraine disability using elements of the PedMIDAS and an Internet headache diary. Cephalalgia. 2014 Apr;34(4):298-306. doi: 10.1177/0333102413508240. Epub 2013 Oct 14. PMID 24126944
- [Background] Heyer GL, Merison K, Rose SC, Perkins SQ, Lee JM, Stewart WC. PedMIDAS-based scoring underestimates migraine disability on non-school days. Headache. 2014 Jun;54(6):1048-53. doi: 10.1111/head.12327. Epub 2014 Apr 7. PMID 24708311
- [Background] Livingston RD, Shockey D, Morton L, Rao S. Pediatric Headache Management and Use of the PedMIDAS. J Dr Nurs Pract. 2019 Apr 1;12(1):24-30. doi: 10.1891/2380-9418.12.1.24. Epub 2019 May 9. PMID 32745052
- [Background] Houts CR, Wirth RJ, McGinley JS, Gwaltney C, Kassel E, Snapinn S, Cady R. Content Validity of HIT-6 as a Measure of Headache Impact in People With Migraine: A Narrative Review. Headache. 2020 Jan;60(1):28-39. doi: 10.1111/head.13701. Epub 2019 Dec 6. PMID 31811654
- [Background] Hershey AD, Powers SW, Vockell AL, LeCates S, Kabbouche MA, Maynard MK. PedMIDAS: development of a questionnaire to assess disability of migraines in children. Neurology. 2001 Dec 11;57(11):2034-9. doi: 10.1212/wnl.57.11.2034. PMID 11739822
- [Background] Genizi J, Lahoud D, Cohen R. Migraine abortive treatment in children and adolescents in Israel. Sci Rep. 2022 May 6;12(1):7418. doi: 10.1038/s41598-022-11467-3. PMID 35523834